CLINICAL TRIAL: NCT05635903
Title: Can Continuous or Intermittent Normal Saline Nebulisation Via a Vibrating Mesh Nebuliser or Intermittent Normal Saline Via a Standard Jet Nebuliser Improve the Lung Physiology and Secretion Viscosity in Mechanically Ventilated Patients?
Brief Title: Jet or Vibrating Mesh Nebulisation for Secretion Management in ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Aerogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN18RM440
Record Dates: First submitted 2022-10-19; First posted 2022-12-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Respiratory Failure; Critical Illness
Keywords: nebuliser; secretions
MeSH Terms: conditions — Respiratory Insufficiency; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continuous nebulisation 0.9% saline Aerogen Solo vibrating mesh Nebuliser (Experimental): Continuous nebulization of 0.9% normal saline using the Aerogen Solo Nebuliser (50mls/24h continuous infusion using a syringe pump)
  Interventions: Procedure: Continuous nebulisation 0.9% saline Aerogen Solo vibrating mesh Nebuliser
- Intermittent nebulisation 0.9% saline Aerogen Solo vibrating mesh Nebuliser (Experimental): Intermittent nebulization of 0.9% normal saline using the Aerogen Solo Nebuliser (5mls 0.9% normal saline nebulised every 6 hours)
  Interventions: Procedure: Intermittent nebulisation 0.9% saline Aerogen vibrating mesh Solo Nebuliser
- Intermittent standard nebulisation of 0.9% saline Intersurgical Cirrus 2 self sealing Jet Nebuliser (Active Comparator): Intermittent standard nebulization of 0.9% normal saline using the Intersurgical Cirrus 2 self-sealing Jet Nebuliser ((5mls 0.9% normal saline nebulised every 6 hours)
  Interventions: Procedure: Intermittent standard intermittent nebulisation of 0.9% saline Intersurgical Cirrus 2 self sealing Jet Nebuliser

INTERVENTIONS:
Procedure: Continuous nebulisation 0.9% saline Aerogen Solo vibrating mesh Nebuliser — Continuous nebulisation of 0.9% saline using the Aerogen Solo vibrating mesh nebuliser
  Arms: Continuous nebulisation 0.9% saline Aerogen Solo vibrating mesh Nebuliser
Procedure: Intermittent nebulisation 0.9% saline Aerogen vibrating mesh Solo Nebuliser — Intermittent nebulisation of 0.9% saline using the Aerogen Solo vibrating mesh nebuliser
  Arms: Intermittent nebulisation 0.9% saline Aerogen Solo vibrating mesh Nebuliser
Procedure: Intermittent standard intermittent nebulisation of 0.9% saline Intersurgical Cirrus 2 self sealing Jet Nebuliser — standard intermittent nebulisation of 0.9% saline using the Intersurgical Cirrus 2 self-sealing Jet Nebuliser
  Arms: Intermittent standard nebulisation of 0.9% saline Intersurgical Cirrus 2 self sealing Jet Nebuliser

SUMMARY:
Critically unwell patients in Intensive Care have a decreased ability to effectively clear secretions. High secretion load is a major risk factor in the failure of tracheal extubation failure and the requirement for reintubation. Extubation failure is a predictor of poor outcome independent of the severity of the underlying illness. Nebulisation of isotonic saline can be employed to manage secretions by reducing the secretion viscosity and facilitating clearance of respiratory sections during tracheal suction.

Standard jet nebulisers have been the mainstay of respiratory section management therapy in critical care since the early 1990s. A more recent development has been the vibrating mesh nebuliser. There is evidence of improved humidification and reduced water particle size and theoretically better transfer to the distal airways.

DETAILED DESCRIPTION:
1.2 Rationale The vibrating mesh nebuliser (Aerogen technology) may be superior to standard nebuliser technology.

1.3 Study hypothesis Improved secretion management with reduced tenacity of respiratory sections and potentially improved lung physiology secondary to improved humidification or reduced size of nebulised particles? 2. STUDY OBJECTIVES

Primary Endpoint Pourability of respiratory secretions (As assessed by the Qualitative Sputum Assessment Tool)

(The QSA score will assess quantity, quality/stickiness/density and colour/appearance of secretions and is described and validated in the literature3,4)

Secondary endpoints

* Volume of secretions (increased or decreased may be beneficial)
* Work of breathing
* Airway resistance
* Number of number of additional nebulised doses of saline or other drugs administered during the study period
* Ease of sampling, in the opinion of treating nurse
* Frequency of requiring changing the HME(heat and moisture exchange) filter
* Length of time on ventilator
* Length of stay in ICU/HDU(Intensive care unit/high dependancy unit)
* ICU Mortality

  3. STUDY DESIGN 3.1 Study Population

A total of 60 patients will be recruited to the study. Each patient will be randomised to receive:

Continuous nebulisation of 0.9% normal saline using the Aerogen Solo Nebuliser (50mls/24h via a syringe feed set) OR

Intermittent nebulisation of 0.9% normal saline using the Aerogen Solo Nebuliser (5mls, 6 hourly) OR

Intermittent standard nebulisation of 0.9% normal saline using the Intersurgical Cirrus 2 self-sealing Jet Nebuliser (5 mls, 6 hourly)

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18-80 years at time of recruitment to study
* Ventilated via an endotracheal tube or tracheostomy with an HME filter in the circuit
* Secretion load defined as patient requiring suctioning at least 2 times in the 6 hours prior to recruitment
* Sputum viscosity with grades 1 to 3 pourability in the Qualitative Sputum Assessment tool
* Not yet received saline nebulisation in the 6 hours prior to recruitment
* Likely to be ventilated via an endotracheal tube or tracheostomy for at least 3 days in the opinion of the treating clinician

Exclusion Criteria:

* Pregnancy
* Pulmonary embolus
* Heart Failure (NYHA Grade III/IV)
* Clinical evidence of frank pulmonary oedema
* Cardiovascular instability (systolic BP ≤75 or heart rate ≥140)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-22 (Actual); Primary Completion 2023-12-22 (Estimated); Study Completion 2023-12-22 (Estimated)

PRIMARY OUTCOMES:
Pourability of respiratory secretions (The QSA score will assess quantity, quality/stickiness/density and colour/appearance of secretions and is described and validated in the literature3,4) | At 1000 and 1600 for 3 days
  Pourability of respiratory secretions as assessed by the QSA (Qualitative Sputum Assessment) Tool 0-4. . As the QSA Tool score ranges from 1 to 4 in increments of 0.5, with 1 being the most pourable and 4 the least pourable.
  (The QSA score will assess quantity, quality/stickiness/density and colour/appearance of secretions and is described and validated Lopez-Vidriero MT, Charman J, Keal E, De Silva DJ, Reid L. Sputum viscosity: correlation with chemical and clinical features in chronic bronchitis. Thorax. 1973 Jul;28(4):401-8. PubMed ID: 4741442

SECONDARY OUTCOMES:
Volume of secretions | At 1000 and 1600 for 3 days
  Total volume in ml of secretions aspirated from the patient's airway at 1000 and 1600 each day
Work of breathing | At 1000 and 1600 for 3 days
  Recorded by ventilator as pressure over volume curve for each breath in joules/min
Airway resistance | At 1000 and 1600 for 3 days
  Recorded by the ventilator in cm H2O/L/sec at 1000 and 1600 each day
Number of number of additional nebulised doses of saline or other drugs administered during the study period | Number of administer nebulised drugs per 24hour per
  Number of nebulized drug doses of drugs administered excluding study drugs
Ease of sampling, in the opinion of the treating nurse | At 1000 and 1600 for 3 days
  Qualitative assessment scale 1-10 . 1 very easy to sample-10 very difficult to obtain a sputum sample.
Frequency of requiring changing the HME filter | Number of filters used in each 24 hour period for 3 days
  Number of HME(heat moisture exchange) filter changes in the previous 24-hour period
Length of time on ventilator | 1 years after admission to ICU/HDU(Intensive care unit/high dependance unit)
  Total number of days ventilated
Length of stay in ICU | Number of day in ICU and HDU at Queen Elizabeth University hospital
  Length of stay in ICU in days
Mortality | 28 days
  Alive at 28 days- Yes/NO

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Sim, MBcHB, Principal Investigator — nhs GGC health board
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thille AW, Richard JC, Brochard L. The decision to extubate in the intensive care unit. Am J Respir Crit Care Med. 2013 Jun 15;187(12):1294-302. doi: 10.1164/rccm.201208-1523CI. PMID 23641924
- [Result] Terzi N, Guerin C, Goncalves MR. What's new in management and clearing of airway secretions in ICU patients? It is time to focus on cough augmentation. Intensive Care Med. 2019 Jun;45(6):865-868. doi: 10.1007/s00134-018-5484-2. Epub 2018 Dec 5. No abstract available. PMID 30519901
- [Result] Jaber S, Quintard H, Cinotti R, Asehnoune K, Arnal JM, Guitton C, Paugam-Burtz C, Abback P, Mekontso Dessap A, Lakhal K, Lasocki S, Plantefeve G, Claud B, Pottecher J, Corne P, Ichai C, Hajjej Z, Molinari N, Chanques G, Papazian L, Azoulay E, De Jong A. Risk factors and outcomes for airway failure versus non-airway failure in the intensive care unit: a multicenter observational study of 1514 extubation procedures. Crit Care. 2018 Sep 23;22(1):236. doi: 10.1186/s13054-018-2150-6. PMID 30243304
- [Result] Keal EE, Reid L. Neuraminic acid content of sputum in chronic bronchitis. Thorax. 1972 Nov;27(6):643-53. doi: 10.1136/thx.27.6.643. PMID 4647626
- [Result] Lopez-Vidriero MT, Charman J, Keal E, De Silva DJ, Reid L. Sputum viscosity: correlation with chemical and clinical features in chronic bronchitis. Thorax. 1973 Jul;28(4):401-8. doi: 10.1136/thx.28.4.401. PMID 4741442
- [Result] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics 2005; 4(4): 287-291.
- [Derived] Arnott A, Hart R, McQueen S, Watson M, Sim M. Prospective randomised unblinded comparison of sputum viscosity for three methods of saline nebulisation in mechanically ventilated patients: A pilot study protocol. PLoS One. 2023 Aug 17;18(8):e0290033. doi: 10.1371/journal.pone.0290033. eCollection 2023. PMID 37590203